CLINICAL TRIAL: NCT03416764
Title: Estradiol-mediated Neural Plasticity as Potential Mediator of Neurofeedback Treatment Change for Traumatized Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0696-17-TLV; TAMC-17-MB-0696-CTIL (Other: TAMC)
Record Dates: First submitted 2018-01-10; First posted 2018-01-31 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD, neurofeedback (NF)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant is aware of treatment group (NF or TAU) Participant is unaware of allocation to treatment estrogen phases (high or low) Investigator and outcome assessor are unaware of group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- EFP-NF (participants without steady menstrual cycle). (Experimental): EFP-NF training, twice a week for a total of 10 sessions .
  Interventions: Device: EFP-NF training
- TAU (No Intervention): Participant will receive no EFP-NF training, and continue their treatment as usual (TAU).
- EFP-NF during HIGH estrogen phase (Experimental): EFP-NF training, twice a week, during high-estrogen phases only (days 7-21 of a 28-day cycle), for a total of 10 sessions.
  Interventions: Device: EFP-NF training
- EFP-NF during LOW estrogen phase (Experimental): EFP-NF training, twice a week, during low-estrogen phases only (days 21-28 of a cycle and days 1-7 of the following cycle,based on a 28-day cycle), for a total of 10 sessions.
  Interventions: Device: EFP-NF training

INTERVENTIONS:
Device: EFP-NF training — Experimental groups (among participants with and without steady menstrual cycle) will receive a total of 10 training sessions during 10 weeks. In addition to EFP-NF training, participants in the experimental groups will continue to be treated as usual at Clinic for Sexual Assault.
  Arms: EFP-NF (participants without steady menstrual cycle).; EFP-NF during HIGH estrogen phase; EFP-NF during LOW estrogen phase

SUMMARY:
Post-traumatic stress disorder (PTSD) is a common debilitating disorder that affects many individuals exposed to aversive events. The severity of PTSD symptoms is positively correlated with amygdala activation. More severe PTSD symptoms following exposure to stressful events, are associated with amygdala hyper-responsivity prior to exposure. A possible intervention for PTSD is Neurofeedback (NF) - a treatment method based on learned self-modulation of neural activity in response to feedback of neural signal. Previous work in our lab established a NF training procedure that utilizes the temporal abilities of EEG with the spatial advantages of fMRI. Further work based on this method using the amygdala BOLD signal (EEG-finger-print, EFP) has demonstrated a potential for improving the ability to self-regulate amygdala activity and to improve emotional regulation in a healthy population. The current study aims to investigate the potential of this method as a therapeutic intervention for PTSD among women with a history of childhood sexual abuse (CSA).

DETAILED DESCRIPTION:
Pretreatment phase- All participants will undergo clinician evaluation, self-report measures and emotional regulation tasks in TASMC. In addition, participants will undergo a functional and structural MRI to characterize brain network responses associated with emotional arousal and regulation.

Participants will be randomized to one of two arms: (1) NF-EFP group and treatment as usual at out-patient clinic (TAU) or (2) TAU (without EFP-NF). If participant has a steady menstrual cycle she will be randomized to one of three arms: (1) NF group administered during low estrogen phase (and maintain TAU); (2) NF group administered during high estrogen phase (and maintain TAU) or (3) TAU (without EFP-NF).

Treatment phase (10 weeks) EFP-NF training, twice a week for a total of 10 sessions. For participants with steady menstrual phase treatment will be administered NF during designated-estrogen phases (high or low).

Treatment as usual: Participants will obtain their regular treatment regimen (pharmacological and psychological) and meet with a psychologist/psychiatrist following the common practice in the clinic.

NF-EFP sessions: For the duration of each NF-EFP session the participant will be seated comfortably in front of a computer screen. A staff member will explain the goal of the meeting to the participant, present the equipment to be used and describe the course of the meeting. The EEG-NF practice will consist of four-minute segments repeated for up to 30 minutes. During each practice segment the participant will be asked to modify visual media that provides feedback on the degree of successful brain training. The duration of one session is approximately 45 minutes.

Post treatment phase -All participants will undergo clinician evaluation, self-report measures and emotional regulation tasks in TASMC. In addition, participants will undergo a functional and structural MRI to characterize brain network responses associated with emotional arousal and regulation.

Follow up- participants will be monitored by self-evaluation questionnaires post treatment.

ELIGIBILITY:
Inclusion Criteria:

Women of age (18-62) :

1. Treated at Clinic for Sexual Assault with stable symptoms.
2. Fulfill screening criteria of DSM-V for PTSD. -

Exclusion Criteria:

1. Pregnancy.
2. Fulfill screening criteria of DSM-V for psychosis.
3. Substance dependence or abuse other than nicotine.
4. Diagnosis of a neurodegenerative disease.
5. Acute illness that could be worsen by the treatment. -

Ages: 18 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-13 (Actual); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Clinical measures- PSTD symptoms | The clinical assessment will be administrated at pre-treatment (baseline) and post-treatment (up to two weeks post-treatment). Additional post-treatment measurements will be administrated at three follow-ups points; 1 month, 3 months and 6 months post
  Change in PTSD symptoms measured by change in Clinician-Administered PTSD Scale (CAPS)

SECONDARY OUTCOMES:
Changes in limbic system connectivity as measured by fMRI | fMRI will be administrated at pre-treatment (baseline) and post-treatment (up to two weeks post-treatment).
  Using fMRI, specific changes in limbic system connectivity will be assessed. Changes in areas in the PFC and limbic regions, all will be measured at post- vs. pre-treatment times
Sleep quality- REM latency and sleep latency | Two nights; first, at pre-treatment (baseline) and second, post-treatment (up to two weeks post-treatment). A post-treatment evaluation will take place within two weeks post treatment (3-3.5 month since the beginning of the study).
  WatchPAT (wearable technology) will track REM latency and sleep latency . These will be compared and corrected using MANOVA as an outcome analysis. To assess sleep globally, we will aggregated: increased sleep latency , reduced sleep efficiency (the ratio of the total time spent asleep compared to the total amount of time spent in bed) and lack of proper deep sleep (quantified using "deep sleep percent" and "REM sleep percent", i.e. the ratio of the total time spent in deep/REM sleep out of the total sleep time) into one reported value. For full explanation and calculation of index see Goldway, et al. (2019).
Emotional regulation choice task | Emotional regulation tasks will be administrated at pre-treatment (baseline) and post-treatment (up to two weeks post-treatment).
  Behavioral - emotional regulation choice task. A computer-based task designed by Sheppes et al. (2011) was used to assess participants'choice between distraction and reappraisal when facing negatively valenced stimuli.
Self-report questionnaires- PCL (PTSD checklist ) | The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).and at three follow-ups points; 1 month, 3 months and 6 months post treatment
  A self-report measure (20 items) of PTSD symptoms reflecting the diagnostic criteria of DSM 4+5. The self-report rating scale is 0-4 for each symptom, Rating scale descriptors are: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) is obtained by summing the scores for each of the items, higher values represent more severe PTSD. Symptom cluster severity scores is obtained by summing the scores for the items within a given cluster, i.e. for DSM 5: cluster B (items 1-5), cluster C (items 6-7), cluster D (items 8-14), and cluster E (items 15-20).
Self-report questionnaires- Beck Depression Inventory (BDI-II) | The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).and at three follow-ups points; 1 month, 3 months and 6 months post treatment
  A 21 item self-administered inventory of depression symptoms and their respective intensity. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. higher values represent more severe depression.
Self-report questionnaires- State-trait Anxiety Inventory (STAI) | The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).and at three follow-ups points; 1 month, 3 months and 6 months post treatment
  A 20 item self-administered inventory of state and trait anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). SUM of scores is obtained, higher scores indicate greater anxiety.
Self-report questionnaires- Toronto Alexithymia Scale (TAS) | The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).and at three follow-ups points; 1 month, 3 months and 6 months post treatment
  20 items self-administered composing the alexithymia scale. The TAS-20 has 3 sub-scales: Difficulty Describing Feelings subscale is used to measure difficulty describing emotions. Difficulty Identifying Feeling subscale is used to measure difficulty identifying emotions. Externally-Oriented Thinking subscale is used to measure the tendency of individuals to focus their attention externally. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. Higher scores represent higher alexithymia rate.
Self-report questionnaires- Dissociative Experience Scale (DES) | The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).and at three follow-ups points; 1 month, 3 months and 6 months post treatment
  28-item self-administered measure of frequency of dissociative experiences. higher DES scores indicate higher dissociative rates.
Self-report questionnaires- Locus of Control (LOC) | The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).and at three follow-ups points; 1 month, 3 months and 6 months post treatment
  24 items self-administered questionnaire intended to measure internal versus external locus of control
Emotional regulation stroop task | Emotional regulation tasks will be administrated at pre-treatment (baseline) and post-treatment (up to two weeks post-treatment).
  emotional Stroop- emotional regulation task, participants viewed fearful or happy facial expressions with superimposed congruent or incongruent words (happy\fear) and were asked to identify the emotional expression while ignoring the words.

CONTACTS AND LOCATIONS:
Overall Officials: Miki Bloch, M.D., Principal Investigator — TASMC Israel
Locations (1):
- Tel Aviv Sourasky Medical Center Tel Aviv, Israel, Tel Aviv, Israel